CLINICAL TRIAL: NCT06177431
Title: An Open Label Extension Study to Investigate the Long Term Safety, Tolerability And Efficacy of Oral Monepantel in Individuals With Motor Neurone Disease Who Previously Completed Study MON-2021-001
Brief Title: An Open Label Extension Study of Monepantel in Individuals With Motor Neurone Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurizon Therapeutics Limited (Industry)
Collaborators: Calvary Health Care Bethlehem (Unknown); Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MON-2023-001
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Motor Neuron Disease
MeSH Terms: conditions — Motor Neuron Disease | interventions — monepantel

STUDY DESIGN:
Intervention Model Description: Open Label Extension
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Monepantel treatment arm (Experimental): Daily dose of 10 mg/kg body weight (QD)
  Interventions: Drug: Monepantel

INTERVENTIONS:
Drug: Monepantel — Monepantel is provided to individuals living with ALS/MND as a white oval tablet to be administered once a day following meals

SUMMARY:
This study is a multicenter, 12-month open label extension study, following Phase 1 Study MON-2021-001, with a single dose of monepantel (MPL) once daily (QD) for the treatment of individuals with MND.

DETAILED DESCRIPTION:
ALS/MND is a progressive, fatal neurodegenerative disease; characterized by motor neuron loss resulting in muscle weakness and atrophy, disability, and eventually death from failure of the ventilatory muscles. The median age of onset is 55 years and average survival is 3-5 years after onset of the first symptoms. The only FDA-approved disease modifying medications confer only a modest survival benefit. Given the poor prognosis and dearth of effective treatments, clinical studies are of primary importance for people with ALS/MND.

Abnormal protein accumulation within motor neurons of the brain associates with the cause of ALS/MND. Inhibition of the mTOR signaling pathway slows disease progression in certain preclinical models of ALS/MND and is suggested to provide synergy with the ALS/MND standard-of-care drug, riluzole. PharmAust has shown that MPL and its major metabolite MPL sulfone (MPLS) have activity against mTOR signaling pathways in humans; based on published data, the inhibition of mTOR may be relevant to the treatment of ALS/MND.

This Phase I Open Label Extension will further test the hypotheses that MPL administration to individuals living with ALS/MND will safely reduce disease associated protein accumulation in motor neurons and provide therapeutic benefit. The safety and tolerability of oral monepantel administration and markers of efficacy will continue to be tested in the same participants that completed the Phase I Study (MON-2021-001).

A daily dose of 10 mg/kg monepantel (QD) will be studied in the Open Label Extension Study (MON-2023-001) to further evaluate long-term safety and efficacy in participants with MND/ALS that completed the Phase I Study (MON-2021-001). Based on the previous pre-clinical efficacy data and clinical safety data, a dose of 10 mg/kg QD is estimated to produce the most robust mTOR inhibition while still being well tolerated. The 10 mg/kg QD dose was the maximum dose evaluated in the Phase 1 Study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to initiation of any study specific procedures and treatment.
2. Individuals who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Able to swallow study drug tablets.
4. Individuals must have completed Study MON-2021-001 and, in the opinion of the investigator, have been compliant with the study procedures and study treatment.
5. Diagnosis of ALS/MND defined as clinically possible, probable, or definite according to Awaji-shima Consensus Recommendations.
6. Not taking riluzole or on a stable dose of riluzole for at least 4 weeks prior to the screening visit; subjects are not allowed to start taking riluzole during the study.
7. Individual has a competent caregiver/support person who can and will be able to support the individual's participation in the study, including assisting with the administration of study drug.
8. Adequate bone marrow reserve, renal and liver function:

   * absolute neutrophil count ≥ 1500/µl.
   * platelet count ≥ 120,000/µl.
   * hemoglobin ≥ 11 g/dL.
   * creatinine clearance ≥ 60 mL/min (Cockroft & Gault formula).
   * alanine aminotransferase and/or aspartate aminotransferase ≤ 3 x upper limit of normal.
   * total bilirubin ≤ 2.0 x ULN.
   * serum albumin ≥ 2.8 g/dL.
9. Women and men with partners of childbearing potential must use effective contraception while on study treatment and women of childbearing potential must be non-lactating.

Exclusion Criteria:

1. Inability to swallow oral medications or presence of a gastrointestinal disorder (e.g., malabsorption) deemed to jeopardize intestinal absorption of study drug.
2. Participated in another investigational drug research study within 4 weeks (28 days) of the Baseline Visit or five half-lives of the drug, whichever is longer.
3. Any other significant illness or condition that in the opinion of the study investigator would interfere with the study conduct.
4. Dementia that may affect either outcome measures or subject understanding and/or compliance with study requirements and procedures.
5. Women and men of childbearing potential not using effective contraception while on study treatment.
6. Women who are breast feeding.
7. Individuals at risk of or are known to carry a SOD1 mutation or VCP mutation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Long-term safety and tolerability | From Baseline to End of Treatment, up to 12 months.
  Assess long-term safety and tolerability of 10 mg/kg body weight (BW) once daily (QD) of monepantel in individuals with Motor Neurone Disease (MND)

SECONDARY OUTCOMES:
Treatment-related changes in serum neurofilament light (NfL) chain levels | From Baseline to End of Treatment, up to 12 months.
  Serum NfL chain levels correlate with disease progression, so stable NfL levels would correlate with stable disease (pg/ml)
Treatment-related changes in urinary p75 levels | From Baseline to End of Treatment, up to 12 months.
  Urinary p75 level reflect nerve damage and therefore increased levels would act as a proxy to disease progression (ng/mg creatinine)
Treatment-related changes on the ALS Functional Rating Scale (ALSFRS) | From Baseline to End of Treatment, up to 12 months.
  The ALS Functional Rating Scale (ALSFRS) is a validated rating instrument for monitoring the progression of disability in patients with amyotrophic lateral sclerosis (ALS). Measurements include: (1) speech (2) salivation (3) swallowing (4) handwriting (5) cutting food and handling utensils (with or without gastrostomy) (6) dressing and hygiene (7) turning in bed and adjusting bed clothes (8) walking (9) climbing stairs and (10) breathing. Possible scores range from 0 (normal function) to 4 (severe loss of function). Change = (Week 4 score - Baseline score)
Treatment-related changes on the Edinburgh Cognitive and Behavioural Amyotrophic Lateral Sclerosis Screen (ECAS) | From Baseline to End of Treatment, up to 12 months.
  The ECAS-cognitive screen is a validated screen comprises 16 items organized into two sub-scales. An ALS-specific sub-scale taps into the cognitive domains of language, verbal fluency, and executive and social functions. A non-ALS-specific sub-scale specifically assesses memory and visuospatial function. The sub-scales of the ECAS-cognitive screen range, respectively, from 0 to 100 and from 0 to 36. Low scores indicate a greater deficit. Change = (Week 4 score - Baseline score)
Treatment-related changes in slow vital capacity (in participants with the capacity to undergo testing) | From Baseline to End of Treatment, up to 12 months.
  A decline in SVC would indicate a decline in respiratory function and is an important indicator of any clinical progression (L/s)
Treatment-related changes in Quality of Life (QOL) Assessment: ALSSQOL-R | From Baseline to End of Treatment, up to 12 months.
  ALSSQOL-R is a 50-item disease-specific questionnaire. Each item is rated on a 10-point Likert scale, with 0 being the least desirable situation and 10 being the most desirable. The instrument produces a single-item QoL score and six domain scores (negative emotion, interaction with people and environment, intimacy, religiosity, physical symptoms, and bulbar function). The ALSSQOL-R is used as QoL outcomes measure to examine the effects of experimental treatments on individual's QoL.
Treatment-related changes in central spinal fluid (CSF) neurofilament light (NfL) chain levels | From Baseline to End of Treatment, up to 12 months.
  CSF NfL chain levels correlate with disease progression. Levels in individuals living with MND are 5 to 10-fold higher than those of healthy individuals (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Mathers, BSc, MB ChB, MRCP(UK), FRACP, Principal Investigator — Calvary Health Care Bethlehem; Dominic Rowe, AM, BSc(Med), MBBS(Hons), PhD, Principal Investigator — Macquarie University, Sydney
Locations (2):
- Australia (2):
  - Macquarie University, Sydney, New South Wales
  - Calvary Health Care Bethlehem, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No